CLINICAL TRIAL: NCT01114360
Title: Melatonin and Nighttime Blood Pressure in African Americans- 8 mg Study
Brief Title: Melatonin and Nighttime Blood Pressure in African Americans-8 mg Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Frederic Rahbari-Oskoui, MD, MSCR, Associate Professor of Medicine, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00021300; 1R21AT004509-01A2 (NIH)
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
Keywords: Melatonin; Hypertension; Blood Pressure; Cardiovascular; Sleep; Nighttime; Nocturnal; Catecholamines; Sympathetic Nervous System; Endothelial function; African American
MeSH Terms: conditions — Hypertension | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Active Comparator): African-American subjects with mild to moderate essential hypertension will be given 8mg time release melatonin for 4 weeks. (either before or after placebo exposure).
  Interventions: Drug: Melatonin; Drug: Placebo
- Placebo (Placebo Comparator): African-American subjects with mild to moderate essential hypertension will be given placebo for 4 weeks (either before or after exposure to melatonin)
  Interventions: Drug: Melatonin; Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Melatonin (N-acetyl-5-methoxytryptamine) is an indoleamine compound. Subjects will receive 8 mg time-release melatonin pills, orally, once per night for 4 weeks.
Drug: Placebo — Subjects received placebo pills (3 pills of 8 mg each) to be taken orally once per night for 4 weeks.

SUMMARY:
This purpose of this study is to test the effect of oral melatonin supplementation (8 mg per night for 4 weeks) on nighttime blood pressure in African Americans with a history of elevated nighttime blood pressure.

DETAILED DESCRIPTION:
The main outcome of interest is the mean nighttime blood pressure. The investigator is also trying to see the mechanism of action of melatonin on blood pressure by analyzing data from sleep studies to see if melatonin lowers blood pressure by providing a better quality of sleep or is that independent of the quality of sleep.

The investigator is also looking into the effect of melatonin on sympathetic nervous system by measuring urinary catecholamines.

Finally, the investigator is looking into changes in vascular biology markers (P-selectin and e-selectin) on melatonin.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 18 to 64
* Prior history of elevated nighttime blood pressure (BP) ((systolic blood pressure (SBP) >115 mmHg))
* Taking no more than 2 antihypertensive medications
* African-American race (self-defined by the participant)

Exclusion Criteria:

* Secondary forms of hypertension
* Presence of other diseases requiring treatment with BP lowering medications
* Known cardiovascular disease (including history of angina pectoris, heart failure, presence of a cardiac pacemaker, history of myocardial infarction or revascularization procedure, or cerebrovascular disease, including stroke and transient ischemic attacks)
* Diabetes mellitus (type 1 or 2)
* Cancer/Malignancy other than nonmelanoma skin cancer
* Primary renal disease
* Serum creatinine > 1.5 mg/dL in men or > 1.4mg/dL in women
* Severe anemia
* Liver enzymes > 2.5 times upper limits of normal
* Hepatitis B, Hepatitis C, or HIV positive as assessed by questionnaire
* Current treatment with or regular use of calcium channel blocking agents, cyclooxygenase-2 or COX2-inhibitors, oral contraceptives, estrogen, sildenafil, vardenafil, tadalafil, antidepressants, corticosteroids, or warfarin
* Current use of melatonin or any sleep aids containing melatonin.
* Regular consumption (1 or more times per week) of any of the following of Vitamin methyl B12, St. Johns Wort, Feverfew, black and white mustard seeds, wolf berry seed
* Severe Sleep apnea
* Night work
* Women who are pregnant, breast-feeding, attempting conception, or planning to attempt conception over the next 6 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic F Rahbari Oskoui, MD, MSCR, Principal Investigator — Emory University; Arlene Chapman, M.D., Principal Investigator — Emory University; Donald Bliwise, Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 patients were screened. 43 patients stopped study participation prior to randomization either due to screen failure or because the decided not to pursue the study procedures.
  37 patients were randomized. There was 1 dropout, and 36 patients completed both arms of the study.
Pre-assignment Details: After signing the ICF and going through screening procedures, 43 patients stopped study participation prior to randomization either due to screen failure or because the decided not to pursue the study procedures.
Groups:
- Placebo/Melatonin: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8mg of placebo for 4 weeks first, followed by 8 mg of time-released melatonin for 4 weeks.
- Melatonin/Placebo: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8 mg of time released melatonin at bed time for 4 weeks, followed by 8 mg of placebo at bedtime for an additional 4 weeks.
Period: Intervention 1 (4 Weeks)
Arm/Group | Placebo/Melatonin | Melatonin/Placebo
Started | 18 | 19
Completed | 18 | 18
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Intervention 2 (4 Weeks)
Arm/Group | Placebo/Melatonin | Melatonin/Placebo
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8mg of time release melatonin or placebo for the first 4 weeks and were then switched to receive either placebo or 8mg of time release melatonin for an additional 4 weeks without any wash out period in between.
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Nighttime Systolic Blood Pressure (SBP)
Description: The nighttime systolic blood pressure (SBP) was recorded using an ambulatory blood pressure (ABP) monitor. The measurements occurring from the onset of self-reported sleep to the end of self-reported sleep were recorded. Means of multiple measurements were reported.
Time Frame: At the end of 4 weeks
Population: 37 subjects enrolled the study. 1 subject did not complete the two arms of the study. 36 subjects completed the study in a crossover design, being their own controls.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Melatonin: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8mg time release melatonin for 4 weeks (either before or after 4 weeks of exposure to placebo).
- Placebo: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received placebo for four weeks (either before or after 4 weeks of exposure to 8 mg daily dose of time release melatonin).
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
mmHg | 126.6 (2.4) | 125.3 (2.5)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; The null hypothesis is that there is no interaction between the order of randomization and primary outcomes; Test type: Superiority or Other; p = 0.075, ANOVA; Two-way repeated measures mixed model ANOVA
Statistical Analysis 2: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.75, ANOVA

2. Secondary Outcome: Mean Nighttime Mean Arterial Pressure (MAP)
Description: Nighttime mean arterial pressure (MAP) is the average blood pressure in the subject's arteries during one cardiac cycle (one complete heartbeat) at night. It is calculated using the formula, MAP = 1/3(SBP-DBP)+DBP; where SBP is the systolic blood pressure and DBP is the diastolic blood pressure. Means of multiple measurements were reported
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
mmHg | 92.9 (1.9) | 92.6 (2.0)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.79, ANOVA

3. Secondary Outcome: Mean Nighttime Heart Rate (HR)
Description: Nighttime heart rate is number of pulsations of the heart per unit of time during nighttime sleep. It is measured in beats per minute (bpm). Ambulatory blood pressure monitoring was used to calculate the heart rate. Means of multiple measurements were reported
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
beats per minute | 75.4 (2) | 76.2 (2.1)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.21, ANOVA

4. Secondary Outcome: Mean Daytime Systolic Blood Pressure (SBP)
Description: The daytime systolic blood pressure was calculated as the average systolic blood pressure during daytime period based on 24hour ambulatory blood pressure monitoring. Means of multiple measurements were reported
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
mmHg | 135.13 (2.2) | 133.9 (2.2)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.64, ANOVA

5. Secondary Outcome: Mean Daytime Diastolic Blood Pressure (DBP)
Description: The daytime diastolic blood pressure was calculated as the average diastolic blood pressure during the daytime period based on 24 hour ambulatory blood pressure monitoring. Means of multiple measurements were reported
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Melatonin: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8mg time release melatonin for 4 weeks (either before or after exposure to 4 weeks of placebo).
- Placebo: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received placebo for four weeks either before or after 4 weeks of exposure to 8mg daily dose of time release melatonin).
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
mmHg | 85.7 (1.6) | 86.2 (1.7)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.89, ANOVA

6. Secondary Outcome: Mean Daytime Mean Arterial Pressure (MAP)
Description: Daytime mean arterial pressure (MAP) is the average blood pressure in the subject's arteries during one cardiac cycle (one complete heartbeat) during the day. It is calculated using the formula, MAP = 1/3(SBP-DBP)+DBP; where SBP is the systolic blood pressure and DBP is the diastolic blood pressure. Means of multiple measurements were reported.
Time Frame: At the end of 4 weeks
Population: 40 subjects enrolled the study. 4 subjects did not complete the study. 36 subjects completed the study in a crossover design, being their own controls.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Melatonin: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8mg time release melatonin for 4 weeks (either before or after 4 weeks of exposure placebo).
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
mmHg | 102.2 (1.7) | 102.1 (1.8)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.97, ANOVA

7. Secondary Outcome: Mean Daytime Heart Rate (HR)
Description: Daytime heart rate is the number of the pulsations of the heart per unit of time during the day. It is measured in beats per minute (bpm). Ambulatory blood pressure monitoring was used to calculate the heart rate. Means of multiple measurements were reported
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
beats per minute | 81 (1.9) | 84.6 (1.9)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.01, ANOVA

8. Primary Outcome: Mean Nighttime Diastolic Blood Pressure (DBP)
Description: The nighttime diastolic blood pressure (DBP) was recorded using an ambulatory blood pressure (ABP) monitor. The measurements occurring from the onset of self-reported sleep to the end of self-reported sleep were recorded. Means of multiple measurements were reported
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
mmHg | 76 (1.7) | 76.2 (1.8)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; The null hypothesis is that there is no interaction between the order of randomization and primary outcomes; Test type: Superiority or Other; p = 0.75, ANOVA

9. Secondary Outcome: Urinary Dopamine Excretion Rate
Description: The rate of urinary dopamine excretion was measured by the Enzyme-Linked Immunosorbent Assay (ELISA) method from urine samples collected overnight.
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml/min
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
ng/ml/min | 140.9 (13.2) | 137.8 (13.0)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.71, Friedman

10. Secondary Outcome: Urinary Noradrenaline Excretion Rate
Description: The rate of urinary noradrenaline excretion was measured by the Enzyme-Linked Immunosorbent Assay (ELISA) method from urine samples collected overnight.
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml/min
Groups:
- Placebo: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received placebo for four weeks ((either before or after 4 weeks of exposure to 8 mg daily dose of time release melatonin).
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
ng/ml/min | 17.5 (3.0) | 19.0 (3.0)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.38, Friedman

11. Secondary Outcome: Urinary Adrenaline Excretion Rate
Description: The rate of urinary adrenaline excretion was measured by the Enzyme-Linked Immunosorbent Assay (ELISA) method from urine samples collected overnight.
Time Frame: At the end of 4 weeks
Population: 40 patients were enrolled in the study. 4 subjects did not complete the study. 36 patients completed the study and were their own controls.
Measure: Mean (Standard Error); unit: ng/ml/min
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
ng/ml/min | 2.75 (0.6) | 2.02 (0.6)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.11, Friedman

12. Secondary Outcome: Plasma E-Selectin
Description: E-Selectin is a marker of endothelial function. Levels of e-selectin were measured from stored plasma using enzyme-linked immunosorbent assay (ELISA).
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Placebo: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received placebo for four weeks (either before or after 4 weeks of exposure to 8mg time release melatonin).
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
ng/ml | 38.6 (2.1) | 38.9 (2.1)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.96, ANOVA

13. Secondary Outcome: Plasma P-Selectin
Description: P-Selectin is a marker of endothelial function. Levels of p-selectin were measured from stored plasma using enzyme-linked immunosorbent assay (ELISA).
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Melatonin: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8mg time release melatonin for 4 weeks (either before or after 4 weeks of placebo) in a crossover design.
- Placebo: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received placebo for four weeks (either before or after exposure to 8mg time release melatonin for 4 weeks).
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
ng/ml | 97.02 (7.6) | 82.7 (7.6)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.25, ANOVA

14. Secondary Outcome: Total Sleep Time
Description: The total sleep time will be measured by polysomnography (PSG) using an Embla polysomnograph. The nocturnal total sleep time (TST) or the the total number of minutes in any stage of sleep during the major nocturnal sleep period was measured by PSG.
Time Frame: At the end of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Groups:
- Melatonin: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8mg time release melatonin for 4 weeks followed by 4 weeks of placebo.
- Placebo: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received placebo for four weeks followed by 8mg time release melatonin for 4 weeks.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
minutes | 399.8 (11.0) | 412.2 (11.1)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Test type: Superiority or Other; p = 0.52, ANOVA

15. Secondary Outcome: Nocturnal Dipping of Blood Pressure
Description: Nocturnal dipping is the mean nighttime to mean daytime systolic and diastolic blood pressure ratios, or the percentage drop in nocturnal SBP compared to day time SBP. Night was defined as 10:00 PM through 5:59 AM. This ratio is calculated by the ambulatory blood pressure readings.
Time Frame: At the end of 4 weeks
Measure: Mean (Standard Error); unit: percentage ratio in night/day SBP
Groups:
- Melatonin; Placebo: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8mg of time release melatonin or placebo for the first 4 weeks and were then switched to receive either placebo or 8mg of time release melatonin for an additional 4 weeks without any wash out period in between.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
percentage ratio in night/day SBP | 5.6 (1.23) | 6.14 (1.30)

16. Secondary Outcome: Percentage of Participants With Melatonin-related Side Effect.
Time Frame: After 4 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of total number of patients
Groups:
- Melatonin: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received 8mg time release melatonin for 4 weeks (either before or after 4 weeks of treatment with placebo).
  Patients were their own controls (cross over design). 40 subjects were randomized to each of the two study arms (total=40). 4 subjects did not complete the study.
- Placebo: African American subjects with mild to moderate essential hypertension and an elevated nighttime blood pressure >115 mmHg received placebo for four weeks (either before or after 4 weeks of treatment with melatonin).
  Patients were their own controls (cross over design). 40 subjects were randomized to each of the two study arms (total=40). 4 subjects did not complete the study.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 36 | 36
percentage of total number of patients | 47.2 | 50

ADVERSE EVENTS:
Time Frame: 4 weeks on each arm.
Arm/Group | Melatonin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 17/36 | 18/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Melatonin (N=36) | Placebo (N=36)
Fatigue (General disorders) | 11 | 13
Daytime drowsiness (General disorders) | 11 | 12
Early Morning Wakening (General disorders) | 12 | 11
Dizziness (General disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 3 | 5
Weakness (General disorders) | 2 | 5
Blurred vision (Eye disorders) | 3 | 4
Heart palpitations (Cardiac disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes